CLINICAL TRIAL: NCT06261879
Title: Non-invasive Biomarker Discovery for Pre-cervical or/and Cervical Cancer--ACTN4 and Other Biomarkers in Menstrual Blood
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: WomenX Biotech Limited (Industry)
Responsible Party: Principal Investigator, Pui Wah Choi, Founder, Principal Investigator, Director, WomenX Biotech Limited
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2023-001
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Cervical Cancer; CIN
Keywords: pre-cervical cancer; cervical cancer; CIN; Sanitary pad; non-invasive detection method; pap smear test
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A sanitary pad as a menstrual blood collector (Experimental): The sanitary pad is similar to the normal sanitary pad.
  Interventions: Device: Special sanitary pad

INTERVENTIONS:
Device: Special sanitary pad — The special sanitary pad is similar to the normal sanitary pad with 0.01 agar gel only. The agar gel is an approved source of food.

SUMMARY:
The goal of this clinical trial is

1. To test the sensitivity and specificity of using ACTN4 from menstrual blood for the detection of pre-cervical or/and cervical cancer.
2. If ACTN4 is not a promising biomarker, other biomarkers will be explored.
3. To develop an effective and non-invasive detection method for pre-cervical or/and cervical cancer.

in Women with menstruation.

The main question it aims to answer is:

To validate whether menstrual blood could be used as a non-invasive means for the detection of pre-cervical or cervical cancer

Participants will

1. Join the briefing session of the study
2. Sign the consent form and health questionnaire
3. Submit the cervical medical report(s) within 3 months or perform sponsored pap smear test
4. Collect the menstrual blood sample

If there is a comparison group: Researchers will compare The diseased group and the healthy group according to the medical reports they provided to see if ACTN4 from menstrual blood is a promising biomarker for the detection of pre-cervical or cervical cancer

DETAILED DESCRIPTION:
First stage of study: Female subjects within the age group will first attend an online research briefing session. After the online briefing session, the participant is provided an opportunity to join a private 1-to-1 consultation session, which enables the participant to be more familiar with the details of the research content, consent form, study procedures, and data confidentiality. If they have no further questions regarding the research content, consent form, etc. during the consultation session. They will sign the consent for participating in the study, they will fill in a questionnaire (attached) and clinic pap smear application form (attached). The questionnaire helps the research team to understand the subject's medical, gynaecological, and sexual histories; a unique identifier code will be given to each subject.

Second Stage of study: The research team will select the subjects based on the questionnaire answers. If the selected subjects have undergone pap test/ HPV test or coloscopy recently, within 3 months, they will submit the related medical record with the unique identifier number to us. If the selected subjects have not undergone pap test/ HPV test or coloscopy recently, within 3 months, they will be sponsored to Pap test or/and HPV genotyping or/and colposcopy at the designated hospitals or clinics. When their Pap test or/and HPV genotyping or/and colposcopy results are available, they or the designated hospitals/ clinics will send us the related medical reports with the unique identifier number.

Third Stage of Study: The participants will be further selected according to the medical records submitted. If the participants were selected to enter the third stage of the study, the selected subjects will submit their menstrual blood to us with a unique identifier number given.

ELIGIBILITY:
Inclusion Criteria:

* Female aged between 18 to 65
* Have menstruation
* Had sex before
* Can read and write Chinese/ English
* Without taking any medication (Except nutritional supplements, traditional Chinese medicine, and health care products etc.)

Exclusion Criteria:

* Subjects who used medication will be excluded from the sample collection. Moreover, subjects with visible signs of gynarcological infections (e.g. gonorrhea, trichomonas vaginalis) or suffered an HIV/ hepatitis B virus (HBV)-infection will be excluded.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
ACTN4 is a promising biomarkers for the detection of pre-cervical/ cervical cancer | From enrollment to sample analysis, 1month
  Hemoglobin will be depleted from samples using NTA agarose beads according to the method of Ringrose and following the manufacturer's instructions [1]. A human ACTN4 ELISA kit (Cusabio Biotech Co. LTD) will be used according to the manufacturer's instructions for revealing the concentration of ACTN4 in the samples [2].
  1. Ringrose, J.H., et al., Highly efficient depletion strategy for the two most abundant erythrocyte soluble proteins improves proteome coverage dramatically. J Proteome Res, 2008. 7(7): p. 3060-3.
  2. ELISA Protocol-Cusabio. Cusabio Life Science-Your Biology Science Partner. 2020 Jul 22; Available from:
  https://www.cusabio.com/m-264.html.

CONTACTS AND LOCATIONS:
Locations (1):
- WomenX Biotech Limited, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Teame H, Addissie A, Ayele W, Hirpa S, Gebremariam A, Gebreheat G, Jemal A. Factors associated with cervical precancerous lesions among women screened for cervical cancer in Addis Ababa, Ethiopia: A case control study. PLoS One. 2018 Jan 19;13(1):e0191506. doi: 10.1371/journal.pone.0191506. eCollection 2018. PMID 29352278
- [Background] Aoki ES, Yin R, Li K, Bhatla N, Singhal S, Ocviyanti D, Saika K, Suh M, Kim M, Termrungruanglert W. National screening programs for cervical cancer in Asian countries. J Gynecol Oncol. 2020 May;31(3):e55. doi: 10.3802/jgo.2020.31.e55. Epub 2020 Feb 26. PMID 32266804
- [Background] Wang B, He M, Chao A, Engelgau MM, Saraiya M, Wang L, Wang L. Cervical Cancer Screening Among Adult Women in China, 2010. Oncologist. 2015 Jun;20(6):627-34. doi: 10.1634/theoncologist.2014-0303. Epub 2015 May 8. PMID 25956407
- See also: Cervical Cancer — https://www.who.int/health-topics/cervical-cancer
- See also: Cervical Cancer: Statistics — https://www.cancer.net/cancer-types/cervical-cancer/statistics.
- See also: Cervical Cancer: Screening and Prevention. Doctor-Approved Patient Information from ASCO — https://www.cancer.net/cancer-types/cervical-cancer/screening-and-prevention.